CLINICAL TRIAL: NCT06182059
Title: Enhanced Recovery After Surgery and Total Knee Replacement: A Prospective, Randomized Study on the Rule of Peripheral Nerve Blocks on Persistent Postoperative Pain Six Months After Surgery
Brief Title: Persistent Post Surgical Pain After Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico di Monza SpA (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, MD, Policlinico di Monza SpA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPSP PTG
Record Dates: First submitted 2023-12-05; First posted 2023-12-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Knee Arthropathy
Keywords: knee arthroplasty; acute postoperative pain; persistent post surgical pain; regional anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fast track (Active Comparator): continuous adductor canal block and ipack block
  Interventions: Procedure: continuous peripheral nerve block
- traditional (Experimental): continuous femoral nerve block and continuous sciatic block
  Interventions: Procedure: continuous peripheral nerve block

INTERVENTIONS:
Procedure: continuous peripheral nerve block — continuous regional anesthesia in total knee replacement

SUMMARY:
Patients undergone total knee replacement are randomized to receive a "fast track" regional anesthesia protocol or a "traditional" regional anesthesia continuous infusion by both a femoral and sciatic catheter to assess if this latter technique may reduce persistent postoperative pain six months after surgery

DETAILED DESCRIPTION:
Patients undergone to primary total knee replacement with spinal anesthesia are randomized to receive a continuous adductor canal block infusion + an ipack block or a continuous femoral nerve block + a continuous sciatic nerve block just at the end of surgery. Both group will receive a multimodal analgesia with paracetamol, ketorolac, desametasone and morphine as a rescue.

ELIGIBILITY:
Inclusion Criteria:

* primary total knee replacement with a written informed consent

Exclusion Criteria:

* Allergy to local anesthetics or any drugs involve in the study
* Controindication to regional anesthesia
* chronic use of opioids
* BMI > 35 kg m2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Persistent post surgical pain | 0-6-month
  Numeric rating score (0-10) over 4 at the follow up 6-month after total knee replacement

SECONDARY OUTCOMES:
acute postoperative pain | 0-72 hours
  Numeric rating score (0-10) over 4 in POD0, POD1, POD2, POD3
Morphine requirement | 0-72 hours
  total morphine administration via PCA in POD0, POD1, POD2, POD3

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico di Monza SPA, Monza, Monza Brianza, Italy